CLINICAL TRIAL: NCT03153449
Title: Multi-Center Clinical Evaluation of the ATTUNE Revision System in Complex Primary Total Knee Arthroplasty
Brief Title: ATTUNE® Revision- Complex Primary in Total Knee Arthroplasty Population
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSJ-2016-03
Record Dates: First submitted 2017-05-07; First posted 2017-05-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Primary Knee Arthroplasty
Keywords: complex primary, deformity, ligamentous laxity
MeSH Terms: conditions — Congenital Abnormalities; Joint Instability | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ATTUNE Revision knee system (Other): The ATTUNE Revision knees system is complementary to the ATTUNE primary knee portfolio and includes both rotating platform (RP) and fixed bearing (FB) configurations. The system includes a full compliment of implants designed to address the challenges faced in complex primary knee surgeries. These implants include Stemmable tibial and femoral components, augments, sleeves and offsets
  Interventions: Device: ATTUNE Revision Knee System in Total Knee Arthroplasty

INTERVENTIONS:
Device: ATTUNE Revision Knee System in Total Knee Arthroplasty — Implants from the ATTUNE Revision Knee System will be used to treat subjects whose surgeons have determined their anatomy is such that the use of revision components are required to perform primary total knee arthroplasty
  Other Names: complex primary knee arthroplasty

SUMMARY:
Five-year, Prospective, multi-center, non-randomized, non-controlled study of the ATTUNE® Revision total knee prostheses, utilizing the fixed bearing (FB) and rotating platform (RP) tibial component with the posterior stabilizing (PS) femoral component in complex primary total knee arthroplasty.

DETAILED DESCRIPTION:
Within primary TKA, there are factors that lead to more complex procedures that include patients with high BMIs, advanced preoperative deformities and ligamentous laxity. Such cases may require the surgeon to treat using ancillary components, such as stems and/or augments and/or additional constraint.

This post-market study will evaluate the short/medium term clinical performance and medium term survivorship of the ATTUNE Revision system system, which includes instrumentation, in complex primary TKA. The study is designed as a worldwide non-comparative, multi-center study with each site initially having a cohort of approximately 20 Subjects to recruit. The study will enroll approximately 200 fixed bearing and approximately 200 rotating platform configurations.

The 2-year KOOS-ADL (activities of daily living) was selected as the primary endpoint because it will evaluate the post-operative period during which outcomes typically plateau and will therefore provide a good indication of longer term outcomes

Male and female Subjects, age 22-80 years, inclusive, who require a primary knee arthroplasty in a joint that, due to deformity, instability, bone loss etc., necessitates the use of implants found within the ATTUNE Revision knee system and are suitable candidates for TKA using the ATTUNE® Revision system are eligible for enrollment in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female and between the ages of 22 and 80 years at the time of consent, inclusive.
2. The decision to have knee replacement with the study device is regardless of the research.
3. The devices are to be used according to the approved indications.
4. Subject that is willing to give voluntary, written informed consent to participate in this clinical investigation and authorize the transfer of his/her information to the Sponsor
5. Subject is currently not bedridden.
6. Subject, in the opinion of the Investigator, is able to understand this clinical investigation and is willing and able to perform all study procedures and follow-up visits and co-operate with investigational procedures.
7. Subject is able to read, and comprehend the Informed Consent Document as well as complete the required PROMs in either English or one of the available translations.
8. Subject has not been diagnosed with an inflammatory arthritis (including gout, rheumatoid, psoriatic etc.)

Exclusion Criteria:

1. The Subject is a woman who is pregnant or lactating.
2. Contralateral knee has already been enrolled in this study. If the Investigator plans to treat a potential study subject with either simultaneous (two (2) knees in one (1) surgical setting) or staged bilateral TKA, then this subject may be enrolled; however, only the first knee may be enrolled into this study.
3. Subject had a contralateral amputation.
4. Previous partial knee replacement (unicompartmental, bicompartmental or patellofemoral joint replacement) or primary TKA in affected knee.
5. Subject is currently diagnosed with radicular pain from the spine that radiates into the limb to receive TKA.
6. Subject has participated in a clinical investigation with an investigational product (drug or device) in the last three (3) months.
7. Subject is currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
8. Subject, in the opinion of the Investigator, is a drug or alcohol abuser (in the last 5 years) or has a psychological disorder that could affect his/her ability to complete patient reported questionnaires or be compliant with follow-up requirements.
9. Subject was diagnosed and is taking prescription medications to treat a muscular disorder that limits mobility due to severe stiffness and pain such as fibromyalgia or polymyalgia.
10. Subject has a significant neurological or musculoskeletal disorder(s) or disease that may adversely affect gait or weight bearing activities (e.g., muscular dystrophy, multiple sclerosis, Charcot disease).
11. Subject has a medical condition with less than five (5) years life expectancy as determined by the Investigator.
12. Subject has been diagnosed with an inflammatory arthritis (including uncontrolled gout, rheumatoid, psoriatic etc.).

    -

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
KOOS ADL | 2 Years
  Evaluate change from preoperative baseline to the 2 yr timepoint in patient reported functional outcome, KOOS-ADL for the ATTUNE® Revision TKA FB and RP configurations.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score - Activities of Daily Living (KOOS-ADL) | Baseline, 5 Year
  Evaluate change from preoperative baseline to the 5 yr timepoint in functional outcomes as measured using KOOS patient reported outcomes measure (PROM).
Patient's Knee Implant Performance (PKIP) | Baseline, 5 Year
  Evaluate change from preoperative baseline to 5 yr timepoint in functional outcomes, satisfaction and quality of life assessments, as measured using the PKIP patient reported outcome measure
American Knee Society Score | Baseline, 5 Year
  valuate change from preoperative baseline to 5 yr timepoint in functional outcomes assessments, patient satisfaction and expectations and clinical evaluations as measured using the AKS measure
EQ-5D-5L | Baseline, 5 year
  Evaluate change from preoperative baseline to 2 and 5 yr timepoints in functional outcomes and quality of life assessments, as measured using the EQ-5D-5L patient reported outcome measure
VAS Pain Score | Baseline, 5 year
  Evaluate change from preoperative baseline to 5 yr timepoint in patient reported pain severity as measured using a modified VAS Pain Score (discrete numbers rather than a continual scale).
American Knee Society Score | Baseline, 5 year
  Evaluate change from preoperative baseline to the 5 yr timepoint in patient reported satisfaction from the AKS 2011 over time as measured using a Likert scale.
American Knee Society Score (surgeon evaluation) | Baseline, 5 year
  Estimate the change from preoperative baseline to the 5 yr timepoint in clinical outcomes using the 2011 AKS (surgeon evaluation)
Adverse Events | Intraoperative, 6 weeks, 1 yr., 2 yr., 3 yr., 4 yr., 5 yr.
  Evaluate type and frequency of Adverse Events
Readmissions | 6 weeks, 1 yr., 2 yr., 3 yr., 4 yr., 5 yr.
  Evaluate the timing, duration and reason for any readmissions stratified by adverse event type (operative site vs. systemic).
Survivorship | 1, 2, 3, 4 and 5 years
  Evaluate survivorship of the ATTUNE® Revision TKA system for the PS FB and PS RP configurations and the combined PS FB and PS RP configurations using Kaplan-Meier survival analysis at 1, 2, 3, 4 and 5 years.
Frequency of radiolucent line occurrence | 1, 2 and 5 years
  Evaluate ATTUNE® Revision TKA fixation through zonal radiographic analysis of the bone-implant interface at 1, 2 and 5 years after surgery compared to the first postoperative radiographs.
Anatomic Tibiofemoral Alignment | 1, 2 and 5 years
  Evaluate any changes in anatomic tibiofemoral alignment at 1, 2 and 5 yrs compared to the first postoperative radiographs.
Femoral component alignment | 1, 2 and 5 years
  Evaluate any changes in femoral component alignment at 1, 2 and 5 yrs compared to the first postoperative radiographs.
Tibial component alignment | 1, 2 and 5 years
  Evaluate any changes in tibial component alignment at 1, 2 and 5 yrs compared to the first postoperative radiographs.
Restoration of joint line | First post-operative radiograph (1 day)
  Radiographically evaluate the restoration of joint line using the first postoperative radiographs according to the methodology of Figgie.

CONTACTS AND LOCATIONS:
Overall Officials: Grant Jamgochian, Study Director — Sponsor GmbH
Locations (34):
- United States (15):
  - Scripps Clinic Torrey Pines, San Diego, California
  - Colorado Joint Replacement, Denver, Colorado
  - Orthopaedic Center of the Rockies, Fort Collins, Colorado
  - Orthopedic Partners, Niantic, Connecticut
  - Florida Orthopedic Associates, DeLand, Florida
  - Arthroplasty Foundation, Louisville, Kentucky
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Rothman Institute, Egg Harbor, New Jersey
  - UNC Orthopaedics, Chapel Hill, North Carolina
  - OrthoCarolina Hip and Knee Center, Charlotte, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Southern Joint Replacement Institute, Nashville, Tennessee
  - Texas Institute for Hip & Knee Surgery, Austin, Texas
  - Fondren Orthopedic Group, Houston, Texas
- Australia (2):
  - Fremantle Hospital, Fremantle
  - St. John of God Murdoch Hospital, Perth
- Krankenhaus der Barmherzigen Schwestern Linz Betriebsgesellschaft m.b.H., Linz, Austria
- Canada (2):
  - London Health Sciences Centre University Hospital, London, Ontario
  - Concordia Joint Replacement, Winnipeg
- France (2):
  - CHRU La Cavale Blanche, Brest
  - Centre Hospitalier Universitaire de Rennes, Rennes
- Germany (2):
  - Klinik und Poliklinik für Orthopädie und Sportorthopädie am Klinikum rechts der Isar der Technischen Universität Münche, Munich
  - Asklepios Orthopädische Klinik Lindenlohe, Schwandorf in Bayern
- South Infirmary Public Hospital, Cork, Ireland
- University Hospital Maastricht, Maastricht, Netherlands
- Wellington Hospital, Wellington, New Zealand
- United Kingdom (7):
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke
  - Victoria Hospital NHS Fife, Kirkcaldy
  - Chapel Allerton Orthopaedic Centre, Leeds
  - James Cook University Hospital, Middlesbrough
  - The Robert Jones and Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry
  - Nuffield Orthopaedic Centre, Oxford
  - Wrightington Hospital, Wigan

IPD SHARING:
Plan to Share IPD: No